CLINICAL TRIAL: NCT05801484
Title: Continuous Infusion Versus Intermittent Administration of Linezolid - Impact on Clinical Outcome and Adverse Reactions in Critically Ill Patients: a Pharmacokinetic and Pharmacodynamic Prospective Study
Brief Title: Pharmacokinetics and Pharmacodynamics of Linezolid Continuous and Intermittent Administration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cluj Municipal Clinical Hospital (Other)
Collaborators: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Bodolea Constantin, Assoc Prof. Dr., Cluj Municipal Clinical Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3/2022
Record Dates: First submitted 2022-11-15; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Side-effect of Antibiotic; Efficacy; Pharmacokinetics; Critical Illness; Intensive Care Unit ICU
Keywords: continuous infusion; intensive care unit; critically ill; linezolid; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: open, prospective, randomized design, with two groups of patients (group with intermittent administration and group with continuous administration of the same daily dose of linezolid).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linezolid continuous infusion (Experimental): In the intervention arm, Linezolid is administered 600 mg as loading dose as an infusion lasting one hour (flow rate 300 ml/h), followed by continuous infusion of 1200 mg linezolid over 24 hours (flow rate 25 ml/h) which is immediately initiated. The continuous infusion is administered until the end of the treatment.
  Interventions: Other: Linezolid continuous infusion
- Linezolid Intermittent administration (Active Comparator): In the comparator arm, 600 mg dose of Linezolid is administered as one-hour infusion (flow rate 300 ml/h). Two doses at 12-h intervals are infused until the end of the treatment.
  Interventions: Other: Linezolid continuous infusion

INTERVENTIONS:
Other: Linezolid continuous infusion — Continuous infusion of 1200 mg linezolid in 24h, after an initial dose of 600 mg linezolid administered as one hour infusion

SUMMARY:
The purpose of this study is to evaluate the therapeutic efficacy expressed in pharmacokinetic/pharmacodynamic (PK/PD) indices, the clinical response and the risk of adverse reactions following the continuous and intermittent administration of linezolid in critical patients in the Intensive Care Unit.

Subject inclusion criteria:

A minimum of 30 subjects in each group will be included in the study, in accordance with the study inclusion criteria:

* patients hospitalized in the intensive care unit,
* female or male sex,
* age over 18 years,
* linezolid is prescribed by the attending physician, in empirical or targeted treatment

Exclusion criteria:

Patients who have documented severe liver failure (Child-Pugh C score). Patients who refuse to sign the informed consent

DETAILED DESCRIPTION:
The clinical study will be conducted in accordance with the protocol approved by the Ethics Commission of the "I.Haţieganu" University of Medicine and Pharmacy and the Ethics Commission of the Municipal Clinical Hospital, from Cluj-Napoca, in accordance with the rules of good clinical study practice.

The study will take place on the Intensive Care Unit of University Clinical Municipal Hospital from Cluj-Napoca, Romania. The analysis of blood drug concentration will be carried out at University of Medicine and Pharmacy 'Iuliu Hatieganu', Pharmacokinetics and Biopharmacy Laboratory, from Cluj-Napoca, Romania.

The objectives of the study are:

* Determination and the comparison of the pharmacokinetic and pharmacodynamic parameters of linezolid administration following intermittent infusion or continuous infusion, in critically ill patients.
* Determination of the minimum inhibitory concentrations (MIC) for linezolid for the identified bacteria (Staphylococcus aureus, Coagulase-Negative Staphylococcus, Enterococcus spp., Streptococcus pneumoniae).

The study will be conducted in the ICU Department of the Municipal Clinical Hospital in Cluj-Napoca, Romania, following an open, prospective, randomized design, with two groups of patients (group with intermittent infusion and group with continuous infusion of the same daily dose of linezolid). The patients that will be included in each group will be the patients in need of intensive care who are prescribed linezolid by the attending physician, as empirical or targeted therapy.

Given the low light stability of the linezolid solution, the infusion bag will be protected with an opaque cover provided by the manufacturer throughout the infusion period. The administration will be carried out with the help of an infusomate.

The duration of the therapy will be established, for each patient, by the attending physician depending on the type, location and severity of the infection in accordance with the recommendations of the therapeutic guidelines.

Throughout the duration of the study, the subjects will receive the treatment according to the recommendations of the attending physician, regardless of the group they belong to, the only difference between the groups refers to the type of infusion used to administer linezolid.

Blood samples (10 samples) will be taken from each volunteer, according to the following schedule: immediately before the start of the infusion (T0) and at 1, 2, 4, 8, 12, 18, 24, 36, 48 hours from initiation of drug infusion. Then, a single daily sample will be taken until the end of the treatment. Blood samples will be used to determine plasma concentrations of linezolid.

The efficacy and safety of the treatment will be evaluated using clinical and paraclinical data which will be correlated with the pharmacokinetic parameters determined for each type of treatment (continuous infusion or intermittent infusion). The data will be recorded in a case report form without disclosing the identity of the patients (each patient will receive a code at the beginning of the study).

Each subject will be followed until discharge or a maximum of 30 days after initiation of therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in the intensive care unit,
* female or male sex,
* age over 18 years,
* linezolid is prescribed by the attending physician, in empirical treatment or based on the antibiogram.

Exclusion Criteria:

* documented severe liver failure (Child-Pugh C).
* no informed consent signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Linezolid plasmatic concentrations | first 2-14 days (during treatment)
  10 plasmatic concentrations in the first 48h of linezolid treatment, then 1 plasmatic concentration per day until the end of the treatment

SECONDARY OUTCOMES:
Linezolid clinical efficacy | from day 1 to day 30 after therapy initiation
  Number of patients with negative cultures after linezolid treatment. Number of patients with laboratory improvement of leucocytes, c reactive protein, procalcitonin after linezolid treatment
Linezolid adverse reactions | from day 1 to day 30 after therapy initiation
  side effects that are described in the summary of the product that may be seen

OTHER OUTCOMES:
Linezolid drug-drug interactions | from day 1 to day 30 after therapy initiation
  drug-drug interactions that are described in the summary of the product that may be seen
Determination of the minimum inhibitory concentration (MIC) for linezolid for the identified bacteria | from day 1
  The linezolid MIC for the gram positive bacteria identified will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Constantin Bodolea, MD, PhD, Principal Investigator — University Of Medicine and Pharmacy Iuliu Hatieganu, Cluj Napoca; Ligia A Hui, PharmD, Principal Investigator — University Of Medicine and Pharmacy Iuliu Hatieganu, Cluj Napoca; Adina Popa, Prof PharmD, Study Chair — University Of Medicine and Pharmacy Iuliu Hatieganu, Cluj Napoca; Laurian Vlase, Prof, PharmD, Study Chair — University Of Medicine and Pharmacy Iuliu Hatieganu, Cluj Napoca
Locations (1):
- University Clinical Municipal Hospital, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hui LA, Bodolea C, Vlase L, Hiriscau EI, Popa A. Linezolid Administration to Critically Ill Patients: Intermittent or Continuous Infusion? A Systematic Literature Search and Review. Antibiotics (Basel). 2022 Mar 24;11(4):436. doi: 10.3390/antibiotics11040436. PMID 35453188